CLINICAL TRIAL: NCT03848884
Title: Impact of Adherence Education and Monitoring on Community Pharmacy Star Ratings and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20014333
Record Dates: First submitted 2019-02-14; First posted 2019-02-21 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Adherence, Patient
MeSH Terms: conditions — Patient Compliance | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adherence monitoring and education (Experimental)
  Interventions: Behavioral: Adherence monitoring and education

INTERVENTIONS:
Behavioral: Adherence monitoring and education — Standardized medication counseling and education combined with individual patient customized guidance and counseling - administered monthly.

SUMMARY:
Does monthly adherence monitoring and education by a pharmacy resident impact Kroger star ratings, compared to the current standard?

DETAILED DESCRIPTION:
To evaluate if a monthly adherence monitoring and education service impacts the percent of patients adherent to oral diabetes and renin-angiotensin system antagonists (RASA) medications based on star ratings. It will also evaluate patient satisfaction of the adherence monitoring and education service, using a standard questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Patients pre-identified by Kroger analytics in ClinicalQ - Patients with PDC < 80%
3. Patient taking oral diabetes medications and/or RASA medications (ACE-I, ARB, direct renin inhibitor)

Exclusion Criteria:

1. Patients who are enrolled in MedSync or Autorefill program
2. Patients who are lost to follow-up
3. Incomplete/missing documentation of an encounter
4. Prisoners, children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Adherence in oral diabetes medications determined by star ratings | Baseline to 6 months
  Determine change in patients who are adherent to oral diabetes medications, determined by pharmacy star ratings in adherence measures; pharmacy analytics determines the star rating measure (on a scale of 1 to 5 stars, with 5 being the highest) before and after the study. A student t-test will be used to determine if there is a difference.
Adherence in renin-angiotensin system antagonists (RASA) medications determined by star ratings | Baseline to 6 months
  Determine change in patients who are adherent to RASA medications, determined by pharmacy star ratings in adherence measures; pharmacy analytics determines the star rating measure (on a scale of 1 to 5 stars, with 5 being the highest) before and after the study. A student t-test will be used to determine if there is a difference.

SECONDARY OUTCOMES:
Change in proportion of days covered (PDC) | Baseline to 6 months
  Determine change in PDC after monthly follow-up on medication adherence and education; pharmacy analytics determines patient PDC in normal practice. The mean PDC for each patient at the end of the six-month study period will be compared to the baseline using a student t-test.

OTHER OUTCOMES:
Satisfaction with education and monitoring service | 6 months
  "Patient Satisfaction Survey" includes an 8-item 5-point likert scale (Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree) about whether or not the pharmacist provided adequate education to the patient, whether or not the patient feels his/her health benefited from the service, and if the patient would recommend the service. The "Patient Satisfaction Survey" will be analyzed using descriptive statistics to determine how satisfied patients were with the medication adherence monitoring and education service.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Venable Goode, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No